CLINICAL TRIAL: NCT00468169
Title: A Randomized Phase II Trial of Concurrent Chemoradiation With Cetuximab (ERBITUX®), 5 Fluorouracil, Hydroxyurea, and Twice-daily Radiation (CetuxFHX) Versus Cetuximab (ERBITUX®), Cisplatin, and Accelerated Radiation With Concomitant Boost (CetuxPX) After Induction Chemotherapy in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Cetuximab (ERBITUX®) Added to Two Concurrent Chemoradiotherapy Platforms in Locally Advanced Head and Neck Cancer
Acronym: EPIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14401A
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Head and Neck Cancer
Keywords: Cetuximab; Erbitux; locally; advanced; head; neck; cancer; neoplasms; squamous; carcinoma; lymphoepithelioma
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms; Carcinoma | interventions — Cetuximab; Fluorouracil; Hydroxyurea; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: Cetuximab+FHX (Experimental): Cetuximab [250mg/m2 (day 1, weekly x10)] + FHX (5-FU [CI: 600mg/m2/day; days 0-5 (120h total) every other week x5], Hydroxyurea [500 mg PO BID, days 0-5 (=11 doses), every other week x5] and twice-daily radiation [150 cGy per fraction - days 1-5, every other week x5 (70-72 Gy total dose)]). Total duration is 10 weeks.
  Interventions: Drug: Cetuximab; Drug: 5-FU; Drug: Hydroxyurea; Radiation: Twice-daily radiation
- B: Cetuximab + PX (Experimental): Cetuximab [250 mg/m2 (day 1, weekly x7)] + PX (Cisplatin [100mg/m2 (week 1 & 4 on day 1 (or 2))], Accelerated fraction radiotherapy with concomitant boost [AFX-CB (72 Gy/42 F/6 W) (3-D or IMRT based)]). Total duration: 7 weeks.
  Interventions: Drug: Cetuximab; Drug: Cisplatin; Radiation: Accelerated fraction radiotherapy with concomitant boost

INTERVENTIONS:
Drug: Cetuximab — 250mg/m2(day 1, weekly x 10);
  Other Names: Erbitux (R)
Drug: 5-FU — 600 mg/m2/day; days 0-5 (120 h total) every other week x 5
  Arms: A: Cetuximab+FHX
Drug: Hydroxyurea — 500 mg PO BID, days 0-5 every other week x 5
  Arms: A: Cetuximab+FHX
Radiation: Twice-daily radiation — 150 cGy per fraction, days 1-5, every other week x 5 (total duration 10 weeks)
  Arms: A: Cetuximab+FHX
Drug: Cisplatin — 100 mg/m2, week 1 and 4 on day 1 (or 2)
  Arms: B: Cetuximab + PX
Radiation: Accelerated fraction radiotherapy with concomitant boost — 72 Gy/42 F/6 W (3-D or IMRT based). Total duration 7 weeks.
  Arms: B: Cetuximab + PX

SUMMARY:
The main purpose of this study is to explore and compare the efficacy of Cetuximab (ERBITUX®) added to two concurrent chemoradiotherapy platforms of different intensity in locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Stage III and IV head and neck cancer
* Patients with squamous cell carcinoma of unknown primary and suspected origin in the head and neck area
* No prior chemotherapy or radiotherapy
* Prior surgical therapy of incisional or excisional biopsy and organ-sparing procedures only
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Normal organ and marrow function

Exclusion Criteria:

* Unequivocal demonstration of metastatic disease
* Known severe hypersensitivity to drugs used in the study
* Treatment with a non-approved or investigational drug within 30 days before Day 1
* Incomplete healing from previous surgery
* Pregnancy or breast feeding
* Uncontrolled intercurrent illness including
* Patients with clinically significant pulmonary dysfunction, cardiomyopathy, or any history of clinically significant CHF
* Acute hepatitis or known HIV
* Severe baseline neurologic deficits
* Prior therapy which specifically and directly targets the EGFR pathway
* Prior severe infusion reaction to a monoclonal antibody

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-07; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Everett E Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A: Cetuximab+FHX: Cetuximab [250mg/m2 (day 1, weekly x10)] + FHX (5-FU [CI: 600mg/m2/day; days 0-5 (120h total) every other week x5], Hydroxyurea [500 mg PO BID, days 0-5 (=11 doses), every other week x5] and twice-daily radiation [150 cGy per fraction - days 1-5, every other week x5 (70-72 Gy total dose)]). Total duration is 10 weeks.
  Cetuximab: Cetuximab - Arm A:250mg/m2(day 1, weekly x 10); Cetuximab - Arm B:250mg/m2(day 1, weekly x 7)
- B: Cetuximab + PX: Cetuximab [250 mg/m2 (day 1, weekly x7)] + PX (Cisplatin [100mg/m2 (week 1 & 4 on day 1 (or 2))], Accelerated fraction radiotherapy with concomitant boost [AFX-CB (72 Gy/42 F/6 W) (3-D or IMRT based)]). Total duration: 7 weeks.
  Cetuximab: Cetuximab - Arm A:250mg/m2(day 1, weekly x 10); Cetuximab - Arm B:250mg/m2(day 1, weekly x 7)
Period: Overall Study
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Started | 57 | 53
Completed | 56 | 53
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Continuous [Mean (Full Range); unit: years] | 56.1 [41 to 81] | 55.6 [32 to 79] | 55.8 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 49 | 44 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 11 | 22
  White | 44 | 39 | 83
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Kaplan-Meier estimate of PFS at 1 years. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 1 years
Measure: Number (95% Confidence Interval); unit: Probability (%)
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Probability (%) | 87.7 [76.0 to 94.0] | 92.5 [81.1 to 97.1]
Statistical Analysis 1: Comparison: A: Cetuximab+FHX; Test type: Superiority or Other; p = 0.1225, Log Rank — Log-rank test comparing PFS between two treatment arms

2. Primary Outcome: Progression Free Survival (PFS)
Description: Time from randomization until disease progression or death from any cause. Kaplan-Meier estimate of PFS at 2 years. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Probability (%)
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Probability (%) | 82.5 [71.9 to 91.5] | 84.9 [72.1 to 92.2]

3. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization until death from any cause. Kaplan-Meier estimate of OS at 2 years.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Probability (%)
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Probability (%) | 91.2 [80.2 to 96.3] | 94.3 [83.5 to 98.1]

4. Secondary Outcome: Objective Response Rate to Induction
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Post-Induction (8 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Participants
  Complete Response (CR) | 7 | 4
  Partial Response (PR) | 47 | 41
  Stable Disease (SD) | 3 | 7
  Progressive Disease (PD) | 0 | 1

5. Secondary Outcome: Objective Response Rate to CRT
Description: Response to CRT was assessed by determining whether there was evidence of residual disease in the primary site via radiographic and clinical examination.
Time Frame: From date of chemoradiotherapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Participants | 3 | 4

6. Secondary Outcome: Residual Lymph Node Disease
Description: Response to CRT was also assessed by determining if there was evidence of residual lymph node disease by neck dissection, if warranted by the presence of any radiographically large (>1.5 cm) or focally abnormal lymph node.
Time Frame: Up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
Number analyzed (Participants) | 57 | 53
Participants | 2 | 6

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | A: Cetuximab+FHX | B: Cetuximab + PX
All-Cause Mortality (participants affected / at risk) | 14/57 | 9/53
Serious Adverse Events (participants affected / at risk) | 7/57 | 14/53
Other Adverse Events (participants affected / at risk) | 57/57 | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Cetuximab+FHX (N=57) | B: Cetuximab + PX (N=53)
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 2 | 5
Infections and infestations - Other, specify (Infections and infestations) | 4 | 0
Thromboembolic event (Vascular disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
G-tube placement (Metabolism and nutrition disorders) | 1 | 3
Malnourished (Metabolism and nutrition disorders) | 0 | 2
Presyncopal episode (Nervous system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Cetuximab+FHX (N=57) | B: Cetuximab + PX (N=53)
Weight loss (Investigations) | 51 | 37
Neutrophil count decreased (Investigations) | 48 | 45
Hemoglobin increased (Investigations) | 43 | 36
White blood cell decreased (Investigations) | 46 | 47
Platelet count decreased (Investigations) | 13 | 13
Creatinine increased (Investigations) | 6 | 4
Nausea (Gastrointestinal disorders) | 49 | 45
Vomiting (Gastrointestinal disorders) | 27 | 19
Mucositis oral (Gastrointestinal disorders) | 57 | 53
Dermatitis radiation (Injury, poisoning and procedural complications) | 56 | 53
Constipation (Gastrointestinal disorders) | 46 | 40
Fatigue (General disorders) | 56 | 53
Nervous system disorders - Other, specify (Nervous system disorders) | 18 | 20
Fever (General disorders) | 23 | 31
Anorexia (Metabolism and nutrition disorders) | 41 | 39
Alopecia (Skin and subcutaneous tissue disorders) | 50 | 49
Pain (General disorders) | 57 | 53
Diarrhea (Gastrointestinal disorders) | 25 | 20
Infections and infestations - Other, specify (Infections and infestations) | 56 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 56 | 53
Dehydration (Metabolism and nutrition disorders) | 50 | 49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes